CLINICAL TRIAL: NCT00000588
Title: Chelation Therapy of Iron Overload With Oral Pyridoxal Isonicotinoyl Hydrazone
Brief Title: Chelation Therapy of Iron Overload With Pyridoxal Isonicotinoyl Hydrazone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 308; R01HL042814 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Anemia (Iron-Loading); Beta-Thalassemia; Hematologic Diseases; Hemoglobinopathies; Thalassemia; Iron Overload
MeSH Terms: conditions — Anemia; beta-Thalassemia; Hematologic Diseases; Hemoglobinopathies; Thalassemia; Iron Overload | interventions — Chelation Therapy

STUDY DESIGN:
Intervention Model Description: Chronic dose according to condition:
  1. Reducing the body iron burden to near-normal levels in non- transfusion-dependent patients with iron-loading anemias (requires chelate- induced iron excretion of at least 0.10 to 0.20 mg Fe/kg/day);
  2. Maintaining near-normal body iron stores in transfusion-dependent patients who have previously been well-chelated with chronic subcutaneous or intravenous desferrioxamine (requires chelate-induced iron excretion of at least 0.25 to 0.40 mg Fe/kg/day);
  3. Reducing the body iron burden to near-normal levels in iron-loaded, transfusion-dependent patients (requires chelate-induced iron excretion greater than 0.40 mg Fe/kg/day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chronic therapy of PIH according to medical condition (Experimental): Half of overall participants will get one of the following doses according to their medical condition:
  1. Reducing the body iron burden to near-normal levels in non- transfusion-dependent patients with iron-loading anemias (requires chelate- induced iron excretion of at least 0.10 to 0.20 mg Fe/kg/day);
  2. Maintaining near-normal body iron stores in transfusion-dependent patients who have previously been well-chelated with chronic subcutaneous or intravenous desferrioxamine (requires chelate-induced iron excretion of at least 0.25 to 0.40 mg Fe/kg/day);
  3. Reducing the body iron burden to near-normal levels in iron-loaded, transfusion-dependent patients (requires chelate-induced iron excretion greater than 0.40 mg Fe/kg/day).
  Interventions: Drug: Chelation therapy; Other: Placebo
- Placebo (Placebo Comparator): Half of the participants will receive a Placebo:
  1. Non-transfusion-dependent patients
  2. Transfusion-dependent patients
  3. Iron-loaded, transfusion-dependent patients
  Interventions: Drug: Chelation therapy; Other: Placebo

INTERVENTIONS:
Drug: Chelation therapy — After an initial 21 day balance study to demonstrate that a selected dose of PIH produced sufficient iron excretion, patients were begun on chronic therapy. PIH or placebo were given on days 4 to 9 and days 13 to 18 in a randomized, double-blind, cross-over design.
  Other Names: Chronic therapy of Pyridoxal Isonicotinoyl Hydrazone
Other: Placebo — Placebo given at same time points as the Intervetnion for each clinical condition.
  Other Names: Control

SUMMARY:
To demonstrate the safety and effectiveness of orally-administered pyridoxal isonicotinoyl hydrazone (PIH) for the chronic treatment of iron overload.

DETAILED DESCRIPTION:
BACKGROUND:

Iron overload in patients with refractory anemia may be the consequence of repeated blood transfusion, of excessive absorption of dietary iron, or of a combination of both. The body lacks any effective means for the excretion of excess iron and in patients with refractory anemia, an inexorable accumulation of iron contained in transfused red cells or absorbed from the diet eventually exceeds the body's capacity for safe storage. Without treatment, widespread iron-induced damage to the liver, heart, pancreas, and other organs is followed by an early death, most often the result of cardiac failure.

Treatment with a chelating agent capable of sequestering iron and permitting its excretion from the body is the most widely-used therapeutic approach. Desferrioxamine was first introduced 30 years ago and is the only iron-chelating agent now in clinical use. A number of recent studies have shown that regular chelation therapy with desferrioxamine can prevent organ damage and improve survival in transfusion-dependent patients with thalassemia major and other disorders. However, desferrioxamine given orally is poorly absorbed and to be effective must be given by subcutaneous or intravenous infusion using a small portable syringe pump, ideally for 12 hours each day. Compliance with this regimen is frequently poor, particularly in adolescents with thalassemia major who may be at greatest risk for the lethal complications of iron overload. With modern transfusion programs, one of the main threats to life in patients with transfusion-dependent anemias is non-compliance with iron-chelation therapy. Moreover, the cost of desferrioxamine therapy in transfusion-dependent therapy exceeds $10,000 per year, in part because the drug must be isolated from bacterial cultures. Despite the limitations, trials of desferrioxamine have validated iron chelation as a therapeutic approach to iron overload.

PIH was first recognized as an effective iron chelator in vitro in 1979. It is easily produced by the Schiff base condensation of two widely used, inexpensive drugs, vitamin B-6 (pyridoxal) and the antituberculous agent isoniazid. The recent Phase I studies of low-dose PIH in healthy controls and volunteers with iron overload have found no evidence of toxicity while producing an amount of iron excretion that would be clinically useful in the treatment of non-transfusion-dependent patients with iron-loading anemias. The trial should provide evidence that orally-administered PIH can be substituted for chronic subcutaneous infusions of desferrioxamine in the management of iron overload in refractory anemia.

The trial was part of an Institute-initiated study on Iron Overload: Cooley's Anemia and Other Disorders.

DESIGN NARRATIVE:

There were three studies in the Phase II trial. Study 1 demonstrated the safety and effectiveness of oral PIH in reducing the body iron burden to near-normal levels in non-transfusion-dependent patients with iron-loading anemias. Study 2 demonstrated the safety and effectiveness of oral PIH in maintaining near-normal body iron stores in transfusion-dependent patients who had previously been well-chelated with chronic subcutaneous or intravenous desferrioxamine. Study 3 demonstrated safety and effectiveness of oral PIH in reducing the body iron burden to near normal levels in iron-loaded transfusion-dependent patients. Studies 1 and 2 were carried out concurrently. Study 3 began after the methods used in the first two studies documented a sufficient level of iron excretion to permit the iron-loaded transfusion patients to keep pace with ongoing transfusional loading and excrete previous accumulations of iron. After an initial 21 day balance study to demonstrate that a selected dose of PIH produced sufficient iron excretion, patients were begun on chronic therapy. PIH or placebo were given on days 4 to 9 and days 13 to 18 in a randomized, double-blind, cross-over design. Study 4 demonstrated the effectiveness in 21 patients of oral deferiprone in inducing sustained decreases in body iron concentrations compatible with the avoidance of complications from iron overload.

Repeat balance studies were carried out at three months, six months, and thereafter at least annually with hematological and biochemical parameters monitored at weekly intervals for the first month, at biweekly intervals for the next two months, and at least monthly thereafter. Studies were conducted at the Cleveland Metropolitan General Hospital and at Siriraj Hospital in Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting any of the following health conditions and eligible for Chronic PIH Treatment
* Non- transfusion-dependent patients with iron-loading anemias
* Transfusion-dependent patients who have previously been well-chelated with chronic subcutaneous or intravenous desferrioxamine
* Iron-loaded, transfusion-dependent patients
* Ages: 18-75 years old

Exclusion Criteria:

* People who are not eligible for chronic PIH therapy and not meet the medical conditions listed in the Inclusion criteria
* Ages: 17 years old or younger or 76 years old or older

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1989-06-05 (Actual); Primary Completion 1993-03-31 (Actual); Study Completion 1995-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Brittenham, Principal Investigator — Case Western Reserve University

REFERENCES:
- [Background] Brittenham GM. Pyridoxal isonicotinoyl hydrazone. Effective iron chelation after oral administration. Ann N Y Acad Sci. 1990;612:315-26. doi: 10.1111/j.1749-6632.1990.tb24319.x. No abstract available. PMID 2291560
- [Background] Brittenham GM. Pyridoxal isonicotinoyl hydrazone: an effective iron-chelator after oral administration. Semin Hematol. 1990 Apr;27(2):112-6. No abstract available. PMID 2190317
- [Background] Nathan DG. An orally active iron chelator. N Engl J Med. 1995 Apr 6;332(14):953-4. doi: 10.1056/NEJM199504063321411. No abstract available. PMID 7877655
- [Background] Olivieri NF, Brittenham GM, Matsui D, Berkovitch M, Blendis LM, Cameron RG, McClelland RA, Liu PP, Templeton DM, Koren G. Iron-chelation therapy with oral deferiprone in patients with thalassemia major. N Engl J Med. 1995 Apr 6;332(14):918-22. doi: 10.1056/NEJM199504063321404. PMID 7877649